CLINICAL TRIAL: NCT05328895
Title: Transcutaneous Auricular Vagus Nerve Stimulation for Meniere Disease: Randomized Trial Controlled
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation for Meniere Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: taVNS-MD-2022
Record Dates: First submitted 2022-03-15; First posted 2022-04-14 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-03

CONDITIONS: Meniere Disease
Keywords: Meniere Disease; taVNS; RCT
MeSH Terms: conditions — Meniere Disease | interventions — Betahistine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- taVNS group (Experimental): taVNS was applied using a Huatuo stimulator (SDZIIB) developed by Suzhou manufacture of Medical Device and Material. Stimulation parameters was 1 mA of electrical current at a frequency of 30 Hz with pulse duration ≤ 1 ms, for 30min, administered twice daily. The two electrodes were placed on the cymba conchae and concha around the left ear. Participants received betahistine mesylate tablet (Merislon, Eisai Co., Ltd., China) with the treatment of 6 mg 3 times a day.
  Interventions: Other: Transcutaneous Auricular Vagus Nerve Stimulation with Betahistine
- Control Group (Placebo Comparator): tnVNS was applied using a Huatuo stimulator (SDZIIB) developed by Suzhou manufacture of Medical Device and Material. Stimulation parameters was 1 mA of electrical current at a frequency of 30 Hz with pulse duration ≤ 1 ms, for 30min, administered twice daily. The two electrodes were placed on the antihelix around the left ear. Participants received betahistine mesylate tablet (Merislon, Eisai Co., Ltd., China) with the treatment of 6 mg 3 times a day.
  Interventions: Other: Transcutaneous Auricular Vagus Nerve Stimulation with Betahistine

INTERVENTIONS:
Other: Transcutaneous Auricular Vagus Nerve Stimulation with Betahistine — Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) on the left ear was selected and stimulated with electronic acupuncture apparatus (Hwato, SDZ-IIB), with continuous wave, 25 Hz in frequency, 4 to 8 mA in intensity depending on patient's tolerance. The first 3 treatments were conducted in hospital, during which, the patients were trained to use the apparatus under the instruction of research staff. Afterwards, the rest treatments were exerted at home, twice a day, after every breakfast and dinner respectively, 30 min each time. The treatment was given from Monday to Friday a week, totally for 12 weeks.
  Participants received betahistine mesylate tablet (Merislon, Eisai Co., Ltd., China) with the treatment of 6 mg 3 times a day.

SUMMARY:
Objective: To evaluate the effect of Transcutaneous auricular vagus nerve stimulation for the patients Meniere disease. Methods: We enrolled 88 patients at Beijing TongRen Hospital. All treatments were self-administered by the patients at home after training at the hospital. Patients completed questionnaires at baseline and after 4 weeks, 8 weeks, 12 weeks. Tinnitus Handicap Inventory (THI), Dizziness Handicap Inventory (DHI), Pure Tone Audiometry, visual scale of ear stuffiness and SF-36 were performed to evaluate the therapeutic effects. A difference of P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 and Age <=70.
2. Clinical diagnosis of meniere disease.

Exclusion Criteria:

1. History of depression, tumors, thyroid disease, diabetes, cardiac diseases.
2. History of Otorhinolaryngology surgery.
3. Pregnant or lactating women.

Ages: 20 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | Change from Baseline scores of THI at 12-weeks post-therapy.
  The THI is a 25-items, self-reported questionnaire regarding tinnitus handicap in daily life. The questionnaire comprises a 12-item functional subscale, an 8-item emotional subscale, and a 5-item catastrophic subscale. The three answer options are "yes," "sometimes," and "no," with scores of 4, 2, and 0, respectively. The overall score is the sum of 25 items (Range: 0-100). Higher scores equate to greater severity of tinnitus symptoms.
  measure the subjective tinnitus symptoms.
Dizziness Handicap Inventory (DHI) | Change from Baseline scores of DHI at 12-weeks post-therapy.
  The DHI is 25-items self-reported questionnaire that used to evaluate the functional, emotional, and physical impact of dizziness on patients' daily life. Among the overall 25 items of questions, 9 items are emotional related, 9 items are functional related, and 7 items are physical related questions. The three answer options are "yes," "sometimes," and "no," with scores of 4, 2, and 0, respectively. The overall score is the sum of 25 items (Range: 0-100). Higher scores equate to greater severity of dizziness symptoms.
Pure tone thresholds. | Change from Baseline level of Pure tone thresholds at 12-weeks post-therapy.
  The pure tone thresholds was performed in a sound-attenuated, double-walled booth with circumaural headphones (Sennheiser HD 280 for frequencies from 250 to 8000 Hz and Sennheiser HD 200 for frequencies from 8000 to 14000 Hz; Sennheiser, Old Lyme, USA) on a certified and calibrated audiometric system (Interacoustics, Middelfart, Denmark).
  Thresholds were measured using a probe-detection paradigm with pure tones presented for 250 ms at frequencies of 250, 500, 1000, 2000, 4000, 8000 Hz for each ear. To determine the LDL, the volume was set to 75 dB at 1000 Hz and then continuously raised in 5 dB steps (every 5 s) until the subject gave the signal that this volume was uncomfortable. When the volume exceeded 110 dB the test was stopped to prevent any hearing damage.
  The severity of hearing impairment was calculated as mild (20-40 dB), moderate (41-70 dB), severe (71-95 dB) and profound (>95 dB). Normal hearing was defined as pure-tone thresholds less than 20 dB.
Visual analogue scale (VAS) | Change from Baseline scores of VAS of aural fullness at 12-weeks post-therapy.
  The VAS scale of aural fullness consists of a 100 mm straight line with defined endpoints ("no aural fullness" and "worst aural fullness imaginable") on which the patients were asked to mark their experienced aural fullness (results in mm) at the actual time ("VAS now"). The higher VAS score (Range: 0-100) is correlated with a severe aural fullness.

SECONDARY OUTCOMES:
The Short Form Health Survey (SF36) | Change from Baseline scores of SF-36 at 12-weeks post-therapy.
  The Short Form Health Survey (SF36) attempts to represent multidimensional health concepts and measurements of the full range of health states, including levels of well-being and personal evaluations of health. SF36 is used widely to assess physical and mental well-being in social and individual contexts. Eight subscales are derived, referring to 8 health concepts: physical functioning (SF36-PF), role functioning-physical (SF36-RP), bodily pain (SF36-BP), general health (SF36-GH), vitality (SF36-VT), social functioning (SF36-SF), role functioning-emotional (SF36-RE), and mental health (SF36-MH). Each subscale ranges from 0 (worst health) to 100 (best health), and a score of 50 represents the mean score for the population.
Video head impulse test (vHIT) | Change from Baseline number of pathological saccades and values of vHIT at 12-weeks post-therapy.
  vHIT was used to assess the function of all the six SCCs by measuring the gain of the vestibulo-ocular reflex. The instrument comprises an inertial measurement unit to measure movements of the head and an infrared camera to record eye movements. vHIT can calculate the mean gain value (ratio of eye to head velocity) for each of the six SCCs, and also detect covert or overt saccades. During the test, goggles were secured firmly to patients' head to ensure that the goggles did not slip from the face during head movement. Patients sat ~1.5 m in front of a wall on which a visual target was affixed. Before testing, head movement and eye movement were calibrated according to the manufacturer's instructions.
  According to manufacture recommendations, normal gain values are expected to range between 0.80 and 1.20 for horizontal canals, and 0.70-1.20 for vertical canals. Pathological saccades and gain values below the normal range were recorded.
The caloric test | Change from Baseline number of abnormal Unilateral Weakness (UW) at 12-weeks post-therapy.
  The caloric test was employed to evaluate the horizontal semicircular canal (SCC). The patients took supine position and raised their head to 30 degrees with a pillow. The right and left ears of the patients were stimulated with cool air (24°C) and warm air (50°C) by using an air caloric irrigator system (Micromedical Technologies Inc., Chatham, IL, USA) and a Brookler-Grams closed-loop irrigation unit. We used videonystagmography (VNG) (Ulmer Inc. Marseille, France) to record horizontal eye movements during the test. The subjects were perfused four times for 60 s.
  After perfusion, the nystagmus was observed for 60 s. Unilateral Weakness (UW) was calculated using the maximal slow phase eye velocity: UW = | (RC + RW) - (LC + LW) | / (RC + RW +LC + LW) × 100%, where RC = right cool, RW = right warm, LC = left cool, and LW = left warm.
  UW >25% was considered abnormal.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing TongRen Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Wu D, Liu B, Wu Y, Wang Y, Sun J, Yang J, Duan J, Liu G, Cao K, Zhang Y, Rong P. Meniere Disease treated with transcutaneous auricular vagus nerve stimulation combined with betahistine Mesylate: A randomized controlled trial. Brain Stimul. 2023 Nov-Dec;16(6):1576-1584. doi: 10.1016/j.brs.2023.10.003. Epub 2023 Oct 13. PMID 37838094